CLINICAL TRIAL: NCT06609746
Title: The Effect of Low FODMAP (Fermentable, Oligo-, Di-, Mono-saccharides and Polyols) Diet with Thyme on Clinical Symptoms and Quality of Life in Patients with Irritable Bowel Syndrome
Brief Title: Effectiveness of Thyme in the Management of Clinical Symptoms in Patients with Irritable Bowel Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Samira Rastgoo, Principal Investigator, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: IR.SBMU.RETECH.REC.1399.1034
Record Dates: First submitted 2024-09-14; First posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Irritable Bowel Syndrome (IBS)
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — thyme extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Thyme (Experimental): Taking thyme extract capsules with a low FODMAP diet
  Interventions: Dietary Supplement: Thyme extract
- placebo (Placebo Comparator): Taking placebo capsules with a low FODMAP diet
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Thyme extract — Three Gastrolit capsules daily with a low FODMAP diet for 8 weeks
  Other Names: Gastrolit
  Arms: Thyme
Other: Placebo — Placebo capsules daily with a low FODMAP diet for 8 weeks
  Arms: placebo

SUMMARY:
The goal of this clinical trial is to learn if thyme supplement enhances the effects of a low FODAMP diet on reducing clinical symptoms and improving the quality of life of patients with irritable bowel syndrome or not.

The main questions it aims to answer are:

1. Does consumption of thyme reduce the severity score of clinical symptoms in patients with irritable bowel syndrome?
2. Does consumption of thyme increase the quality of life score in patients with irritable bowel syndrome? Researchers will compare thyme supplementation with placebo to see if thyme supplement enhances the effects of a low FODAMP diet on clinical symptoms and quality of life in patients with irritable bowel syndrome.

Participants will:

1. Receive thyme supplement plus a low FODMAP diet or placebo with low FODMAP diet for 8 weeks.
2. Recorde 3 days (1weekend and 2 workday) dietary recalls at week 4 and week 8 to assess adherence to the low FODMP diet.
3. Visit the clinic at the beginning of the study and the end of the study for a check-up and score record

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-65;
* Patients with irritable bowel syndrome;
* Body Mass Index in the range of 18-25 kg/m2

Exclusion Criteria:

* Any organic intestinal disease;
* Medical history of chronic gastrointestinal and colorectal disease;
* Any major bowel surgery;
* Medical history of liver and kidney disorders;
* Regular use of laxative, anti-diarrhea and anti inflammatory medications.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-10-21 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Irritable Bowel Syndrome symptom severity score | baseline and 8 weeks following therapy
  The primary outcome measure will be a change in the Irritable Bowel Symptom Severity Scale (IBS-SS) from baseline to 8 weeks at the conclusion of therapy. The IBS-SS scale ranges from 0 to 500 . Scores of 75-175, 175-300, and 300-500 indicate mild, moderate, and severe cases.

SECONDARY OUTCOMES:
Defecation frequency | baseline and 8 weeks following therapy
  The secondary outcome measure will be a change in stool frequency from baseline to 8 weeks at the conclusion of therapy. Stool frequency (number of stools per day) is assessed through an interview
Stool consistency | baseline and 8 weeks following therapy
  The secondary outcome measure will be a change in stool consistency from baseline to 8 weeks at the conclusion of therapy. Stool consistency is assessed using the validated Bristol Stool Form Scale.
Quality of life score | baseline and 8 weeks following therapy
  The secondary outcome measure will be a change in quality of life from baseline to 8 weeks at the conclusion of therapy. The quality of life (QoL) is assessed by using a self-report QoL measure specific to IBS (IBS-QoL) with 34 items. Each item has a 5-point Likert scale. Items scores are summed to derive the overall score and transformed to a 0- to 100-scale. The higher scores indicate a better QoL.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR